CLINICAL TRIAL: NCT05233332
Title: A Phase Ⅱ, Multicenter Open-label Study to Investigate the Efficacy and Safety of HL-085 Combined With Vemurafenib in Patients With Metastatic Colorectal Cancer (mCRC)
Brief Title: Study of HL-085 and Vemurafinib in Metastatic Colorectal Cancer (mCRC)
Acronym: mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-201
Record Dates: First submitted 2022-01-21; First posted 2022-02-10 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: CRC
Keywords: metastatic colorectal cancer (mCRC); HL-085; Vemurafenib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- phase IIa: HL-085 in Subjects With BRAF V600E-Mutated CRC (Experimental): 12mg BID HL-085
  Interventions: Drug: HL-085
- phase IIa: HL-085+Vemurafenib in Subjects With BRAF V600E-Mutated CRC (Experimental): 12mg BID HL-085+720mg BID Vemurafenib
  Interventions: Drug: HL-085; Drug: Vemurafenib
- phase IIa: HL-085+Vemurafenib in Subjects With RAS or other BRAF-Mutated or MEK1/2-Mutated CRC (Experimental): 12mg BID HL-085+720mg BID Vemurafenib
  Interventions: Drug: HL-085; Drug: Vemurafenib
- phase IIb: HL-085+Vemurafenib in Subjects With BRAF V600E-Mutated CRC (Experimental): 12mg BID HL-085+720mg BID Vemurafenib
  Interventions: Drug: HL-085; Drug: Vemurafenib

INTERVENTIONS:
Drug: HL-085 — 12mg BID HL-085
Drug: Vemurafenib — 720mg BID Vemurafenib
  Other Names: ZELBORAF
  Arms: phase IIa: HL-085+Vemurafenib in Subjects With BRAF V600E-Mutated CRC; phase IIa: HL-085+Vemurafenib in Subjects With RAS or other BRAF-Mutated or MEK1/2-Mutated CRC; phase IIb: HL-085+Vemurafenib in Subjects With BRAF V600E-Mutated CRC

SUMMARY:
The study consists of the two parts, phase IIa and phase IIb.

DETAILED DESCRIPTION:
The study consists of the two parts, phase IIa and phase IIb. Phase IIa study is to assess the safety and the antitumor activity in patients with mCRC and to recommend reasonable dosage regimen of HL-085 for phase IIb study. Phase IIb is a pivotal study to evaluate HL-085 plus Vemurafenib in patients with BRAFV600E mCRC whose disease has progressed after 1 or 2 prior regimens in the metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to enrollment；
* Adults 18 years of age or older, male or female;
* Histologically- or cytologically-confirmed CRC that is metastatic disease, and a) progression of disease or intolerance after line 1 or line 2 therapy，or inappropriate for line 1 therapy (for phase Ⅱa); b) progression of disease or intolerance after line 1 or line 2 therapy (for phase Ⅱb);
* Patient must have measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST version 1.1);
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Life expectancy ≥ 3 months;
* Able to take the medicine orally;
* Adequate bone marrow and organ function.

Exclusion Criteria:

* Prior treatment with any RAS inhibitors, RAF inhibitors, or MEK inhibitors;
* History or screening evidence of retinal diseases;
* Impaired cardiovascular function or clinically significant cardiovascular and cerebrovascular diseases;
* Previous or current neuromuscular diseases that is associated with CK elevation (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy, rhabdomyolysis syndrome);
* Impaired liver function, defined as Child-Pugh Class B or C;
* Toxicity has not recovered to grade 0 or 1 from prior anticancer therapy (except for alopecia, pigmentation, and grade 2 chemotherapy-related neurotoxicity);
* Use of any medications or foods that are strong inhibitors or inducers of cytochrome P450 (CYP) 3A4/5 within 7 days prior to the start of study treatment or during the study period, , drugs with a narrow therapeutic window for CYP1A2 metabolism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
ORR（by investigator） | up to 12 months
  Phase IIa：ORR per the RECIST version 1.1，defined as the number of patients achieving an overall best response of CR or partial response (PR) divided by the total number of patients
ORR（by ICR） | up to 12 months
  Phase Ⅱb：ORR per the RECIST version 1.1，defined as the number of patients achieving an overall best response of CR or partial response (PR) divided by the total number of patients

SECONDARY OUTCOMES:
PFS（by investigator） | up to 12 months
  Phase IIa：PFS，defined as the time from first dose to the earliest documented disease progression or death due to any cause
PFS（by ICR） | up to 12 months
  Phase IIb：PFS，defined as the time from first dose to the earliest documented disease progression or death due to any cause
DOR（by investigator） | up to 12 months
  Phase IIa：DOR，Duration of response is defined as subjects who show a confirmed clinical response (CR) or partial response (PR), the time from first documented evidence of CR or PR until the first documented sign of disease progression or death
DOR（by ICR） | up to 12 months
  Phase IIb：DOR，Duration of response is defined as subjects who show a confirmed clinical response (CR) or partial response (PR), the time from first documented evidence of CR or PR until the first documented sign of disease progression or death
DCR（by investigator） | up to 12 months
  Phase IIa：Proportion of subjects with response defined as CR, PR, and SD throughout the study from subjects first dose to disease progression or death
DCR（by ICR） | up to 12 months
  Phase IIb：Proportion of subjects with response defined as CR, PR, and SD throughout the study from subjects first dose to disease progression or death
OS | up to 24 months
  OS is defined as the time from the date of taking drugs to the date of death due to any cause
Number of Adverse Events | up to 12 months
  Number of Treatment-Related Adverse Events as Assessed by CTCAE v5.0 will be counted

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, Ph.D, Study Director — Shanghai Kechow Pharma, Inc.
Locations (1):
- Beijing Oncology Hospital, Beijing, Beijing Municipality, China